CLINICAL TRIAL: NCT04288024
Title: The Learning Effects of Task-priority Strategy on Dual-task Weight Shifting and Brain Plasticity in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201907085RIND
Record Dates: First submitted 2020-02-24; First posted 2020-02-27 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2020-02

CONDITIONS: Postural and Suprapostural Performance During Dual Tasking in Patients With Parkinson's Disease
Keywords: Parkinson; dual-task training; attention; electroencephalogram (EEG)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postural (Experimental): During training, participants in this group are instructed to focus on their posture during weight-shifting.
  Interventions: Behavioral: Weight-shifting training
- Suprapostural (Experimental): During training, participants in this group are instructed to focus on their suprapostural task during weight-shifting.
  Interventions: Behavioral: Weight-shifting training

INTERVENTIONS:
Behavioral: Weight-shifting training — Postural task: Participants are standing with their weak side on the force plate. During the task, they wight-shift from side to side ranging from 10 to 90 percent of their body weight.
  Suprapostural task: Participants hold a tray with their arms beside the body, 90 degrees of elbow flexion. They rotate the tray left and right for 45 degrees respectively.
  During their task, participants should weight-shift and rotate the tray at the same time.

SUMMARY:
(1) postural and suprapostural performance of a dual task would be differently affected by the strategy of task prioritization and (2) the cortical activation is different according to attentional focus strategies.

DETAILED DESCRIPTION:
These hypothesis would be tested by gait performance, suprapostural accuracy and relative power spectrum of EEG.

ELIGIBILITY:
Inclusion Criteria:

* 1. modified H-Y stage II-III Parkinson's disease 2. No other diseases 3. Non-demented PD 4. Non-tremor PD

Exclusion Criteria:

* None

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
EEG relative power in the delta band | 60 minutes
  postural and suprapostural performance of a dual task
EEG relative power in the theta band | 60 minutes
  postural and suprapostural performance of a dual task
EEG relative power in the alpha band | 60 minutes
  postural and suprapostural performance of a dual task
EEG relative power in the beta band | 60 minutes
  postural and suprapostural performance of a dual task
EEG relative power in the gamma band | 60 minutes
  postural and suprapostural performance of a dual task
COP trajectory recorded from the force plate | 60 minutes
  performance of the postural task
Angles from inclinometer | 60 minutes
  performance of the suprapostural task

SECONDARY OUTCOMES:
Gait velocity from GAITRite | 5 minutes
  gait performance
Cadence from GAITRite | 5 minutes
  gait performance
Mean step length from GAITRite | 5 minutes
  gait performance
Step-to-step variability from GAITRite | 5 minutes
  gait performance

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No